CLINICAL TRIAL: NCT05085873
Title: Sodium Oxybate Versus Midazolam for Comfort Sedation
Acronym: ONAMI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020-CHITS-002; 2021-001961-19 (EudraCT Number)
Record Dates: First submitted 2021-09-23; First posted 2021-10-20 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-11

CONDITIONS: Palliative Care
Keywords: Sedation; End-of-life; Palliative care; Midazolam; Sodium oxybate
MeSH Terms: conditions — Death | interventions — Sodium Oxybate; 4-hydroxybutyric acid; Midazolam

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants won't be aware of the sedative treatment administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium oxybate (Experimental)
  Interventions: Drug: Sodium Oxybate injection
- Midazolam (Active Comparator)
  Interventions: Drug: Midazolam injection

INTERVENTIONS:
Drug: Sodium Oxybate injection — * Induction dosage : 60 mg/kg by direct intravenous injection.
  * Continuous dosage : 45 mg/kg/h by continuous intravenous injection.
  * Additional dosage if the Richmond Agitation Sedation Scale (RASS) score exceeds -4 : 1000 mg sodium oxybate by direct intravenous injection bolus every hour at most until RASS score reaches -4.
  Sedation maintained until patient death.
  Other Names: Gamma-Hydroxybutyric acid; 4-hydroxybutanoic acid
  Arms: Sodium oxybate
Drug: Midazolam injection — * Induction dosage : 1 mg every 3 min by direct intravenous injection until RASS score reaches -4 (with a maximum of 30 min).
  * Continuous dosage : Half of titration dosage every hour by continuous intravenous injection.
  * Additional dosage if the RASS score exceeds -4 : 1 mg every 3 min by direct intravenous injection (without exceeding 10 mg/h).
  Sedation maintained until patient death.
  Arms: Midazolam

SUMMARY:
The study aims at deepen the proof level of sodium oxybate use for comfort sedation at the end of life in a palliative care unit by comparing it to midazolam in a prospective randomized study with blinded efficacy evaluation. The study will be carried out for a period of 24 months with a recruitment objective of 22 patients with refractory suffering and with a short-term prognosis.

DETAILED DESCRIPTION:
In certain cases, terminally-ill patients may show persistent symptoms despite numerous efforts to find a comfort treatment without causing impaired consciousness. In these cases and after a collegial discussion, sedation may be offered.

Midazolam is then the most typically used sedative agent. However, it has limitations: frequent awakenings, tolerance and major respiratory depression. Furthermore, the use of midazolam as a "gold standard" in palliative sedation at the end of life falls under expert consensus without a high level of evidence.

Sodium oxybate (GammaOH®), is an ancient molecule used in anesthesia and other medical fields. It appears to be an attractive alternative to midazolam. Study hypothesis is as follows: deep sedation induced by sodium oxybate (RASS: -4 or -5) is more constant and sustainable than by using midazolam which can cause fluctuating effects and requires frequent dosage adjustments. The single-blind clinical trial aims at comparing the possibility to obtain constant deep sedation using midazolam or sodium oxybate. Before the induction, the patient is not aware of the medication used. The medical team must be aware of it because the two administration procedures are too different.

ELIGIBILITY:
Inclusion Criteria:

* patient hospitalized in a palliative care unit
* patient aged 18 or over
* patient with an estimated vital prognosis of a few hours to a few days*
* patient with persistent suffering despite optimal palliative care*
* patient gave informed consent in advance or if unable to do so, consent given by a family member or legal representative (patients under guardianship)
* patient covered by a social security scheme. * Validated after collegial and multidisciplinary discussion including the opinion of a doctor outside the palliative care team.

Exclusion Criteria:

* contraindication or known allergy to sodium oxybate or midazolam
* significant risk of seizure
* venous access not possible
* pregnancy or breastfeeding
* person in exclusion period from another research protocol at the time of consent signing
* any condition which in the investigator's opinion could increase and jeopardize persons safety in case of research participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Reaching and maintaining a comfort sedation defined by a target RASS score of -4 | From inclusion until death, up to 12 hours
  Treatment is defined as successful when reaching and consistently maintaining the target score; treatment is defined as not successful when not reaching the target score at induction or not maintaining a score of <= -4 for patients who initially reached the target.

SECONDARY OUTCOMES:
Adverse events | From inclusion until death, up to 12 hours
  Number of clinical adverse events recorded in both arms.
Survival time | From inclusion until death, up to 12 hours
  Time span between induction of sedation and death.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François CIAIS, MD, Study Director — Centre Hospitalier Princesse Grace - Monaco
Locations (1):
- Centre Hospitalier Princesse Grace, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ciais JF, Jacquin PH, Pradier C, Castelli-Prieto M, Baudin S, Tremellat F. Using Sodium Oxybate (Gamma Hydroxybutyric Acid) for Deep Sedation at the End of Life. J Palliat Med. 2015 Oct;18(10):822. doi: 10.1089/jpm.2015.0221. Epub 2015 Aug 24. No abstract available. PMID 26302340
- [Result] Ciais JF, Jacquin PH, Gac Marrec A, Decorbez A, Saudemont G, Dugourd C, Berthier F, Payen D. Sodium oxybate versus midazolam for end-of-life continuous deep sedation: a randomised controlled trial. BMJ Support Palliat Care. 2025 Dec 21:spcare-2025-005747. doi: 10.1136/spcare-2025-005747. Online ahead of print. PMID 41429434